CLINICAL TRIAL: NCT03232866
Title: Effects of Load Monitoring on Pilates Training: a Randomized Clinical Trial
Brief Title: Effects of Load Monitoring on Pilates Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Franciele Marques Vanderle, PhD, Paulista University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69459517.8.0000.5402
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Pilates Method; Exercise
Keywords: Exercise Movement Techniques; Exercise; Monitoring, Physiologic; Heart Rate; Autonomic Nervous System; Heart rate variability
MeSH Terms: conditions — Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): (n = 20) will practice Pilates exercises
  Interventions: Other: Pilates exercise
- Control group (No Intervention): (n = 20) will not carry out the intervention

INTERVENTIONS:
Other: Pilates exercise — Pilates methods exercises
  Arms: Experimental group

SUMMARY:
There has been an increasing awareness about the need to practice some physical activity, including several objectives, mainly as a preventive character. From this perspective, notice the use of the Pilates method as an instrument of therapeutic exercise for the protection and promotion of health. However, despite being popularly performed, there is still no scientific evidence on the standardization of the use of the method and its progression to an adequate prescription of physical training. The objective is monitoring the progression of loads of a 12-week training among the basic, intermediate and advanced levels of the Pilates method through heart rate (HR), subjective exertion perception (PSE) and heart rate variability (HRV). In addition, analyzing the effect of the method on cardiorespiratory and autonomic parameters. 40 healthy men aged 18-36 will receive Pilates training for 12 weeks. After the initial assessment and familiarization with the method, the training period will begin totalizing 36 sessions for three months, where each class lasts approximately 1 hour. During the three months, the participants must pass through the three levels of training: Basic, Intermediate and Advanced. During each session, the investigators will initially collect: psychological questionnaire, visual analogue pain scale (VAS), and cardiorespiratory parameters (systolic and diastolic blood pressure, HR, respiratory rate and partial oxygen saturation). Throughout the session a heart rate meter will be positioned on the chest of the participant to capture HR, which will occur every five minutes together with the PSE illustrated in the model proposed by Borg. At the end of each session, the cardiorespiratory parameters will be collected again. In addition, cardiorespiratory parameters and HRV will be analyzed at baseline and after three months of training. In the case of HRV analysis, linear methods in the time and frequency domain will be verified. For the statistical analysis of the cardiorespiratory and autonomic parameters in the pre and post training moments will be used paired t test for normal data or Wilcoxon test for non normal data. For the analysis of the training load will be used the correlation of Pearson or Sperman according to normality. The definition of cutoff points for the HRV and PSE indices will be obtained by the ROC curve.

ELIGIBILITY:
Inclusion Criteria:

* male sex
* healthy
* aged between 18 and 36 years

Exclusion Criteria:

* smokers
* alcoholics
* use drugs that influenced cardiac autonomic activity
* cardiovascular, metabolic or endocrine diseases.

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the indices of heart rate variability in different levels of pilates (basic, intermediate and advanced) | Eight (transition from basic to intermediate level) and twelfth week (transition from intermediate to advanced level)

SECONDARY OUTCOMES:
Change from baseline in the subjective perception of effort in different levels of pilates (basic, intermediate and advanced) | Eight (transition from basic to intermediate level) and twelfth week (transition from intermediate to advanced level)
Change from baseline in the heart rate in different levels of pilates (basic, intermediate and advanced) | Eight (transition from basic to intermediate level) and twelfth week (transition from intermediate to advanced level)

CONTACTS AND LOCATIONS:
Locations (1):
- Franciele Marques Vanderlei, Presidente Prudente, São Paulo, Brazil

REFERENCES:
- [Derived] Cavina AP, Silva NM, Biral TM, Lemos LK, Junior EP, Pastre CM, Vanderlei LC, Vanderlei FM. Effects of 12-week Pilates training program on cardiac autonomic modulation: a randomized controlled clinical trial. J Comp Eff Res. 2021 Dec;10(18):1363-1372. doi: 10.2217/cer-2021-0195. Epub 2021 Oct 21. PMID 34672201
- [Derived] de Souza Cavina AP, Pizzo Junior E, Machado AF, Biral TM, Pastre CM, Vanderlei FM. Load monitoring on Pilates training: a study protocol for a randomized clinical trial. Trials. 2019 Oct 17;20(1):597. doi: 10.1186/s13063-019-3684-x. PMID 31623638